CLINICAL TRIAL: NCT06977880
Title: A Phase 1, First-in-human Study of MORF-440 in Healthy Participants, Including Single and Multiple Ascending Dose Cohorts
Brief Title: A Phase 1, First-in-human Study of MORF-440 (LY4292009) in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Morphic Therapeutic, Inc. (A Wholly Owned Subsidiary of Eli Lilly and Company) (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 27728; Morf-440-101 (Other: Eli Lilly and Company); J6O-MC-UMAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-12; First posted 2025-05-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Cohort A1 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort A2 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort A3 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort A4 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort A5 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort A6 (Optional) (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort B1 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort B2 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort B3 (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Cohort B4 (Optional) (Experimental): Participants received LY4292009 orally.
  Interventions: Drug: LY4292009
- Placebo (Placebo Comparator): Participants receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4292009 — Administered orally
  Arms: Cohort A1; Cohort A2; Cohort A3; Cohort A4; Cohort A5; Cohort A6 (Optional); Cohort B1; Cohort B2; Cohort B3; Cohort B4 (Optional)
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending doses of MORF-440 administered to healthy participants single-ascending dose (SAD) and maximum ascending dose (MAD) substudy.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within 18.0 kg/m² to 30.0 kg/m², inclusive
* If male, meets one of the following:

  * can procreate and agree to use one of the accepted to use one of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration.
  * is unable to procreate; defined as surgically sterile (i.e., has undergone a vasectomy at least 180 days prior to the first study drug administration)
* if female, meets one of the following:

  * is of childbearing potential and agrees to use an acceptable contraceptive method.
  * is of non-childbearing potential, defined as either:

    * Surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or
  * is in a postmenopausal state:

    * At least 1 year without menses and without an alternative medical condition prior to the screening, and follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at screening or at least 1 year without menses and without an alternative medical condition prior to the screening, follicle stimulating hormone FSH levels < 40 milli-international units per milliliter (mIU/mL) and estradiol serum level ≤150 picomole/Liter (pmol/L) at screening

Exclusion Criteria:

* Female who is lactating or who is pregnant according to the pregnancy test at screening or prior to the first study drug administration, or planning to become pregnant during the study period up to 30 days after the last study drug administration
* Nicotine intake (e.g., smoking, nicotine patch, nicotine chewing gum, chewing tobacco, electronic cigarettes) within 1 month before screening and/or inability to refrain from nicotine from screening until the end of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Event (SAEs) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | Baseline to Study Completion (Up to Day 17)
Percentage of Participants with TEAEs and SAEs in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | Baseline to Study Completion (Up to Day 7)
Number of Participants with One or More Serious Adverse Event(s) (SAEs) in (Cohort A1-A6) and MAD (Cohort B1-B4) | Baseline to Study Completion (Up to Day 7)
Change from Baseline in Laboratory Parameter and Vital Signs in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | Baseline to Study Completion (Up to Day 7)
Number of Participants with Clinically Significant Changes in Cardiovascular Evaluation in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | Baseline to Study Completion (Up to Day 7)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Maximum observed plasma concentration
PK: Time to Maximum Concentration (Tmax) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Time to reach Cmax, defined as the first point if multiple maximum values occur.
PK: Area Under the Concentration Curve (AUC) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
PK: Time to Half Life (T1/2) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Apparent first-order terminal phase half-life, calculated as 0.693/λ
PK: AUC From Time Zero to Infinity (AUC 0-inf) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Area under the concentration-time curve from time 0 extrapolated to infinity. Calculated as the sum of AUC0-t plus the ratio of the last measurable concentration to the terminal phase rate constant (λz).
PK: CL/F in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Apparent total clearance after oral administration, calculated as Dose/AUC0-inf
PK: Vd/F in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Apparent volume of distribution during terminal phase after oral administration, calculated as Dose/[λz*AUC0-inf]
PK: Urine: Ae(total) in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  otal amount of urinary excretion (cohorts participating in urinary PK sample collection only)
PK: CLR in SAD (Cohort A1-A6) and MAD (Cohort B1-B4) | SAD Cohorts: Predose up to Day 4 Postdose
  Clearance of urinary excretion (cohorts participating in urinary PK sample collection only), calculated as Ae/AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Altasciences Company Inc., Mount Royal, Canada

IPD SHARING:
Plan to Share IPD: No